CLINICAL TRIAL: NCT03851432
Title: Efficacy and Safety of Janagliflozin in Combination With Metformin in Type 2 Diabetes Patients With Inadequate Glycemic Control With Metformin Alone
Brief Title: Janagliflozin Treat Type 2 Diabetes Mellitus (T2DM) Inadequately Controlled With Metformin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5695-DIA-3002
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — janagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Janagliflozin 25 mg plus metformin (Experimental): Each patient will receive 25 mg of Janagliflozin plus metformin for 52 weeks (a 24-week core period followed by a 28-week extension period)
  Interventions: Drug: Janagliflozin plus metformin
- Janagliflozin 50 mg plus metformin (Experimental): Each patient will receive 50 mg of Janagliflozin plus metformin for 52 weeks (a 24-week core period followed by a 28-week extension period)
  Interventions: Drug: Janagliflozin plus metformin
- Placebo/Janagliflozin plus metformin (Placebo Comparator): In the core period, each patient will receive placebo plus metformin for 24 weeks and will then switch from placebo to 25 mg or 50 mg of Janagliflozin plus metformin until Week 52.
  Interventions: Device: Placebo plus metformin

INTERVENTIONS:
Drug: Janagliflozin plus metformin — Janagliflozin: Tablets, Oral, 25 mg, Once daily, 52 weeks The patient's stable dose of background therapy of metformin should be continued throughout the study.
  Arms: Janagliflozin 25 mg plus metformin
Drug: Janagliflozin plus metformin — Janagliflozin: Tablets, Oral, 50 mg, Once daily, 52 weeks The patient's stable dose of background therapy of metformin should be continued throughout the study.
  Arms: Janagliflozin 50 mg plus metformin
Device: Placebo plus metformin — Placebo: Tablets, Oral, 25/50 mg, Once daily, 24 weeks The patient's stable dose of background therapy of metformin should be continued throughout the study.
  Arms: Placebo/Janagliflozin plus metformin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Janagliflozin compared to placebo, both in combination with Metformin, in Chinese patients with type 2 diabetes mellitus (T2DM) inadequately controlled with Metformin alone.

DETAILED DESCRIPTION:
A multicentre, randomized, double-blind, placebo-controlled, parallel-group study (a 24-week core period followed by a 28-week extension period), to evaluate the efficacy and safety of Janagliflozin (25 mg and 50 mg) compared to placebo, all in combination with Metformin, in patients diagnosed with T2DM who are not achieving an adequate response from Metformin monotherapy. Approximately 390 patients with inadequate glycemic control with Metformin monotherapy will receive once-daily double-blind treatment with Janagliflozin 25 mg or 50 mg , both in combination with Metformin , for 52 weeks, or receive 24 weeks of double-blind treatment with placebo in combination with Metformin followed by 28 weeks of single-blind treatment with Janagliflozin 25 mg or 50 mg, both in combination with Metformin. During the treatment, if a patient's glycemic level remains high despite treatment with study drug and reinforcement with diet and exercise, the patient will receive treatment with Linagliptin (rescue therapy) consistent with local prescribing information.

ELIGIBILITY:
Inclusion Criteria:

* T2DM Patients with inadequate glycemic control (HbA1c level≥7.0% and ≤10.5% at baseline) on metformin monotherapy.
* Body Mass Index: 18.0~35.0 kg/m2 (both inclusive)

Exclusion Criteria:

* History of type 1 diabetes mellitus (T1DM), diabetes caused by pancreatic injury, or secondary diabetes (e.g., diabetes caused by Cushing's syndrome or acromegaly)
* More than 10% change in body weight within the 3 months before screening
* Any laboratory test indicators meet the following standards:

  * fasting plasma glucose ≥ 15 mmol/L
  * aspartate aminotransferase, alanine aminotransferase levels > 3 times the upper limit of normal (ULN); total bilirubin > 1.5 times ULN
  * hemoglobin < 100 g/L
  * eGFR < 60 mL/min/1.73m2
  * fasting triglycerides > 5.64 mmol/L (500 mg/dL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) From Baseline to Week 24 (Core period) | Baseline and Week 24
  To examine whether the mean change in HbA1c from Baseline to Week 24 with Janagliflozin is superior to placebo

SECONDARY OUTCOMES:
Change in HbA1c From Baseline to Week 52 | Baseline and Week 52
  To compare the mean change in HbA1c from Baseline to Week 52 between groups
Percentage of Patients With HbA1c <7% at Week 24 (Core period) and Week 52 (Extension period) | Week 24 and week 52
  To compare the percentage of patients with HbA1c <7% at Week 24 (core period) and Week 52 (extension period) between groups
Percentage of Patients With HbA1c <6.5% at Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the percentage of patients with HbA1c <6.5% at week 24 (core period) and Week 52 (extension period) between groups
Change in Fasting Plasma Glucose (FPG) From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in fasting plasma glucose (FPG) from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in 2-hour Post-prandial Glucose From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in 2-hour post-prandial glucose from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Blood Lipids (total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in blood lipids (total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Blood Pressure (systolic blood pressure and diastolic blood pressure) From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in blood pressure (systolic blood pressure and diastolic blood pressure) from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Body Weight From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in body weight from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Fasting C-peptide From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in fasting C-peptide from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Insulin Sensitivity From Baseline to Week 24 (Core period) and Week 52 (Extension period) by calculation Homeostasis model assessment-insulin resistance | Baseline, Week 24 and Week 52
  To compare the mean change in insulin sensitivity from Baseline to Week 24 (core period) and Week 52 (extension period) between group by calculation Homeostasis model assessment-insulin resistance
Change in β-cell Function From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in β-cell function from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Percentage of Patients Who Have Received Rescue Therapy at Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the percentage of patients who have received rescue therapy by Week 24 (core period) and Week 52 (extension period) between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Linong Ji, Beijing, Beijing Municipality, China